CLINICAL TRIAL: NCT03080337
Title: Group Prenatal Care Compared to Traditional Prenatal Care for Women With Pre-gestational Diabetes: A Randomized Clinical Trial.
Brief Title: Group vs. Traditional Diabetes Prenatal Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is being closed prematurely due to resource availability and agreement constraints with the collaborating research site.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-015; A532860 (Other: UW Madison); SMPH/OBSTET & GYNECOL/OBSTET (Other: UW Madison)
Record Dates: First submitted 2017-02-27; First posted 2017-03-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Care (No Intervention): If the participant is randomized to the individual prenatal care model, she will continue to receive individualized care in the prenatal clinic. This includes being seen by both a MFM specialist and possibly an endocrinologist at each prenatal visit. During the prenatal visit, the individual caregivers are responsible for discussing educational topics that they feel are relevant to the patient. Patients are seen every two weeks for Traditional Care.
- Group Care (Experimental): If the participant is randomized into the group prenatal care model she will be placed in a group of approximately 6-10 women of approximately the same gestational age. These women will then have sessions scheduled at the same intervals they would have had their traditional prenatal visits, every two weeks until 36 weeks and then weekly until delivery, 12 sessions in total. Each session will last between 90-120 minutes. In the group prenatal care model, the entire visit time will be face to face with a provider and the group. Billing will be done through the standard reimbursement system since the program will follow the schedule of prenatal visits recommended by the American Congress of Obstetricians and Gynecologist.
  Interventions: Other: Group Care

INTERVENTIONS:
Other: Group Care — Participation in 12 group sessions with 6-10 women who are also pregnant and have diabetes.
  Arms: Group Care

SUMMARY:
This study aims to use an innovative and integrated educational curriculum to deliver prenatal care and diabetes care for pre-gestational diabetic women from approximately the first trimester of pregnancy through delivery and the early postpartum period in a group care model. The group care model will be compared to a control group, a traditional, individual care model.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed viable pregnancy at the time of enrollment.
* Able to provide consent for participation.
* Diabetes diagnosed prior to 12 weeks gestation.
* Initiation of care by 20 weeks gestation.
* Age 18 years or older.

Exclusion Criteria:

* Not planning to deliver at UnityPoint Health- Meriter Hospital.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Compliance with glucose testing over time | 2 years
  Compare the glucose compliance of participants in the group care model to the control group: a traditional, individual care model.

SECONDARY OUTCOMES:
Maternal Weight Gain (kilograms) | 2 years
  Compare maternal weight gain of participants in the group care model to the control group: a traditional, individual care model.
Length of stay for delivery (days) | 2 years
  Compare maternal hospital length of stay for delivery of participants in the group care model to the control group: a traditional, individual care model.
Presence of infection (Y/N) | 2 years
  Compare presence of infection in participants in the group care model to the control group: a traditional, individual care model.
Type of Delivery (Vaginal, C-Section, Vacuum, Forceps, other) | 2 years
  Compare type of delivery in participants in the group care model to the control group: a traditional, individual care model.
Blood Pressure (mm Hg) | 2 years
  Compare blood pressures in participants in the group care model to the control group: a traditional, individual care model.
Neonatal Birth Weight (grams) | 2 years
  Compare neonatal birth weight of participants in the group care model to the control group: a traditional, individual care model.
Neonatal Length of stay (days) | 2 years
  Compare neonatal length of stay of participants in the group care model to the control group: a traditional, individual care model.
Neonatal APGAR Score (0-10) | 2 years
  Compare neonatal APGAR score of participants in the group care model to the control group: a traditional, individual care model.
Gestational Age at Delivery (weeks) | 2 years
  Compare gestational age at delivery of participants in the group care model to the control group: a traditional, individual care model.
Pregnancy related and Diabetes related knowledge acquired during pregnancy (survey) | 2 years
  Compare pregnancy and diabetes related knowledge of participants in the group care model to the control group: a traditional, individual care model.
Patient and care giver satisfaction (survey) | 2 years
  Compare satisfaction of participants and their respective providers in the group care model to the control group: a traditional, individual care model.
Cost-effectiveness (dollars per hour) | 2 years
  Compare cost-effectiveness of the group care model to the control group: a traditional, individual care model.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Hoppe, DO, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UnityPoint Health- Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in a REDCap database with University Hospitals, Cleveland.
Supporting Information: Study Protocol, CSR
Time Frame: At time of study completion for up to 1 year.
Access Criteria: De-identified data variables will be shared as this will be a shared enrollment effort.